CLINICAL TRIAL: NCT01760525
Title: A Phase I, Open-label, Multi-center, Dose Escalation Study of Oral CGM097, a p53/HDM2-interaction Inhibitor, in Adult Patients With Selected Advanced Solid Tumors
Brief Title: A Phase I Dose Escalation Study of CGM097 in Adult Patients With Selected Advanced Solid Tumors
Acronym: CCGM097X2101
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCGM097X2101; 2012-000940-87 (EudraCT Number)
Record Dates: First submitted 2013-01-02; First posted 2013-01-04 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Solid Tumor With p53 Wild Type Status
Keywords: p53, solid tumor
MeSH Terms: interventions — NVP-CGM097

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CGM097 - Dose escalation (Experimental)
  Interventions: Drug: CGM097
- CGM097 - Dose Expansion at MTD or RP2D (Experimental)
  Interventions: Drug: CGM097

INTERVENTIONS:
Drug: CGM097 — Patients treated with CGM097

SUMMARY:
This is a first in human phase I study of single agent CGM097 in patients with advanced solid tumors who have progressed despite standard therapy or for whom no standard therapy exists. The tumor must be characterized by p53wt status. The study consists of a dose escalation part where patients will receive escalating doses of CGM097, and a dose expansion part in which patients are given CGM097 at the maximum tolerated dose (MTD) or Recommended Phase 2 Dose (RP2D). Each dose escalation step will be decided based on the recommendation from an adaptive Bayesian logistic regression model (BLRM).

DETAILED DESCRIPTION:
This is a multi-center, open-label, dose finding, phase I study of single agent CGM097, administered in patients with advanced solid tumors who have progressed despite standard therapy or for whom no standard therapy exists. Patients' tumors must be characterized by p53wt status.

The study consists of a dose escalation part, where cohorts of three to six newly enrolled patients will receive escalating doses of CGM097, and a dose expansion part, in which patients are given CGM097 the maximum tolerated dose (MTD) or Recommended Phase 2 Dose (RP2D). Novartis and the site investigators will jointly decide on each dose escalation step based on the recommendation from an adaptive Bayesian logistic regression model (BLRM). If safety data should indicate a lower increment than suggested by the BLRM, the next dose level (DL) will be adjusted accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Patient has advanced solid malignancy that has progressed despite standard therapy, or for which no effective standard therapy exists
* Tumor of the patient is p53wt
* Evaluable disease as determined by RECIST 1.1
* WHO performance status 0-2

Exclusion criteria:

* Prior treatment with CGM097 or other p53/HDM2-interaction inhibitor
* Patient with symptomatic or growing CNS metastatic lesions
* Concurrent other malignancy
* Clinically significant cardiac disease as defined in the protocol
* Diagnosis of acute or chronic pancreatitis
* Concomitant therapy that precludes enrollment, as defined in the protocol
* Women of child-bearing potential, unless they are using highly effective methods of contraception during dosing and for 2 weeks after study drug discontinuation
* Pregnant or nursing women

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-03-20 (Actual); Primary Completion 2020-07-24 (Actual); Study Completion 2020-07-24 (Actual)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicities | From day 1 to day 28 of treatment
  To characterize the maximum tolerated dose (MTD) and/or identify the recommended dose for expansion(RDE) of CGM097. Dose Limiting Toxicities will be listed and their incidence summarized by primary system organ class, worst grade based on CTCAE version 4.03 and type of Adverse Event

SECONDARY OUTCOMES:
Pharmacokinetic profile of CGM097 | At Cycle 1 Day 1, 2, 5, 8, 15 and 22, then each first day of the Cycle (28 days per Cycle) until discontinuation.
  Plasma concentration of CGM097
Tumor response per RECIST | Baseline, then every third cycle (approximately every 12 weeks), until disease progression or discontinuation.
  This includes duration of response and progression free survival
Pharmacodynamic effect of CGM097 | At baseline, Cycle 2 Day 8 and at disease progression.
  Changes of tumors markers in tumor tissue and blood
Changes in laboratory values, vital signs or cardiac functionality, dose reduction, dose interruption and dose intensity, incidence and severity of adverse events. | At Cycle 1 Day 1, 2, 5, 8, 15, 22 and 28, Cycle 2 Day 1, 8,15 and 22, then each Day 1 and 15 of the Cycle until discontinuation. For dose interruption, dose intensity and adverse events: each day of the Cycle until discontinuation (28 days per Cycle).
  Changes in laboratory values, vital signs or cardiac functionality, dose reduction, dose interruption and dose intensity, incidence and severity of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- Dana Farber Cancer Institute SC (2), Boston, Massachusetts, United States
- Novartis Investigative Site, Lyon, France
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bauer S, Demetri GD, Halilovic E, Dummer R, Meille C, Tan DSW, Guerreiro N, Jullion A, Ferretti S, Jeay S, Van Bree L, Hourcade-Potelleret F, Wuerthner JU, Fabre C, Cassier PA. Pharmacokinetic-pharmacodynamic guided optimisation of dose and schedule of CGM097, an HDM2 inhibitor, in preclinical and clinical studies. Br J Cancer. 2021 Aug;125(5):687-698. doi: 10.1038/s41416-021-01444-4. Epub 2021 Jun 17. PMID 34140638
- See also: Study Results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17833